CLINICAL TRIAL: NCT06269497
Title: TiO2-scaffolds for Alveolar Ridge Preservation
Acronym: TIOSCAFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Jan Eirik Ellingsen, Professor, University of Oslo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018/2300
Record Dates: First submitted 2023-11-30; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Alveolar Bone Resorption
Keywords: Scaffold; Bone resorption
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Intervention Model Description: Observational study / clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scaffold (Experimental): After tooth extraction will one scaffold be placed in the extraction alveola, covered by a membrane and then covered by the gingival tissue.
  Interventions: Procedure: Scaffold placement; Radiation: CBCT

INTERVENTIONS:
Procedure: Scaffold placement — The scaffold is placed in the alveola following extraction
Radiation: CBCT — A Cone Beam Computer Tomography (CBCT) is taken of the area of interest after surgery

SUMMARY:
The goal of this clinical trial is to evaluate the safety of placing TiO2 scaffolds in alveolar ridge and to evaluate if the scaffold material contributes to maintain the anatomy and the volume of the alveolar process after tooth extraction.

DETAILED DESCRIPTION:
The primary objective of the clinical trial is to evaluate the safety of placing TiO2 scaffolds in alveolar ridge.

The secondary objectives are; (1) to assess anatomical changes as measured by intraoral digital scanning at the time of extraction, after 6 months. (2) to evaluate soft tissue inflammation at 1, 2, 4, 12 and 24 weeks post-surgery, (3) to assess the preservation of the alveolar ridge following placement of TiO2 scaffold in the alveolae after tooth extraction, (4) to assess bone mineralization and quantitative healing in bone biopsies obtained at implant installation in the preserved site 6 months following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 20 years, and present with a molar or premolar planned for extraction

Exclusion Criteria:

* Individuals with medical conditions that may affect soft tissue or bone metabolism
* Previous local radiotherapy
* Current use of chemotherapy
* Systemic long-term corticosteroid treatment.
* Diabetes
* Smokers (> 10 cigarettes/day).
* Patients with active of untreated periodontal disease.
* Present or past use of bisphosphonate treatment
* Pregnant or nursing subjects
* > class 2 according to the ASA (American Society of Anesthesiologists) physical status classification
* Acute infection or no apical periodontitis visible on radiograph of tooth planned for extraction.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Adverse reactions | Through study completion, an average of 1 year
  Evaluate and register any adverse reactions following placement of the scaffold

SECONDARY OUTCOMES:
Anatomy | 6 months after surgery
  Evaluate if the anatomy of the alveolar process is maintained or changed, analysis with use of cone-beam-computer-tomography showing the bone at the site immediately after surgery and 6 months after surgery. Any difference in bone volume will be recorded.
Inflammation | Through study completion, an average of 1 year
  Evaluate if any inflammatory response appeared in the surrounding tissues following placement of the scaffold according to the modified Landry index (Pippi 2017), The inflammation parameters are recorded with "yes" or "no" regarding presence.
Mineralization | Evaluation of the histology, specimens tasken 6 months after surgery.
  Evaluate bone ingrowth and mineralization of the pores in the scaffold material by the use of micro-ct analysis, histology and immune histology

CONTACTS AND LOCATIONS:
Overall Officials: Jan Eirik Ellingsen, DDS, PhD, Principal Investigator — University of Oslo
Locations (1):
- Faculty of Dentistry, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muller B, Reseland JE, Haugen HJ, Tiainen H. Cell growth on pore-graded biomimetic TiO2 bone scaffolds. J Biomater Appl. 2015 Apr;29(9):1284-95. doi: 10.1177/0885328214559859. Epub 2014 Nov 13. PMID 25394623
- [Background] Tiainen H, Lyngstadaas SP, Ellingsen JE, Haugen HJ. Ultra-porous titanium oxide scaffold with high compressive strength. J Mater Sci Mater Med. 2010 Oct;21(10):2783-92. doi: 10.1007/s10856-010-4142-1. Epub 2010 Aug 14. PMID 20711636
- [Background] Sabetrasekh R, Tiainen H, Lyngstadaas SP, Reseland J, Haugen H. A novel ultra-porous titanium dioxide ceramic with excellent biocompatibility. J Biomater Appl. 2011 Feb;25(6):559-80. doi: 10.1177/0885328209354925. Epub 2010 Jan 20. PMID 20089606
- [Background] Tiainen H, Wohlfahrt JC, Verket A, Lyngstadaas SP, Haugen HJ. Bone formation in TiO2 bone scaffolds in extraction sockets of minipigs. Acta Biomater. 2012 Jul;8(6):2384-91. doi: 10.1016/j.actbio.2012.02.020. Epub 2012 Mar 3. PMID 22395069
- [Background] Sabetrasekh R, Tiainen H, Reseland JE, Will J, Ellingsen JE, Lyngstadaas SP, Haugen HJ. Impact of trace elements on biocompatibility of titanium scaffolds. Biomed Mater. 2010 Feb;5(1):15003. doi: 10.1088/1748-6041/5/1/015003. Epub 2010 Jan 7. PMID 20057018
- [Background] Tiainen H, Verket A, Haugen HJ, Lyngstadaas SP, Wohlfahrt JC. Dimensional Ridge Preservation with a Novel Highly Porous TiO(2) Scaffold: An Experimental Study in Minipigs. Int J Biomater. 2012;2012:851264. doi: 10.1155/2012/851264. Epub 2012 Oct 3. PMID 23091493
- [Background] Le Thieu MK, Homayouni A, Haeren LR, Tiainen H, Verket A, Ellingsen JE, Ronold HJ, Wohlfahrt JC, Cantalapiedra AG, Munoz FMG, Mendana MP, Lyngstadaas SP, Haugen HJ. Impact of simultaneous placement of implant and block bone graft substitute: an in vivo peri-implant defect model. Biomater Res. 2021 Nov 25;25(1):43. doi: 10.1186/s40824-021-00245-3. PMID 34823602
- [Background] Thieu MKL, Haugen HJ, Sanz-Esporrin J, Sanz M, Lyngstadaas SP, Verket A. Guided bone regeneration of chronic non-contained bone defects using a volume stable porous block TiO2 scaffold: An experimental in vivo study. Clin Oral Implants Res. 2021 Mar;32(3):369-381. doi: 10.1111/clr.13708. Epub 2021 Jan 28. PMID 33420723
- [Background] Thieu MKL, Stoetzel S, Rahmati M, El Khassawna T, Verket A, Sanz-Esporrin J, Sanz M, Ellingsen JE, Haugen HJ. Immunohistochemical comparison of lateral bone augmentation using a synthetic TiO2 block or a xenogeneic graft in chronic alveolar defects. Clin Implant Dent Relat Res. 2023 Feb;25(1):57-67. doi: 10.1111/cid.13143. Epub 2022 Oct 12. PMID 36222116
- [Background] Pippi R. Post-Surgical Clinical Monitoring of Soft Tissue Wound Healing in Periodontal and Implant Surgery. Int J Med Sci. 2017 Jul 18;14(8):721-728. doi: 10.7150/ijms.19727. eCollection 2017. PMID 28824306
- [Derived] Nysaether I, Haugen HJ, El Khassawna T, Jamous R, Afnan S, Santacroce M, Arvidsson LZ, Hildebrand T, Lyngstadaas SP, Ellingsen JE. Clinical Performance of Ultra-Porous TiO2 Scaffold as Bone Graft Substitute in Human Alveolar Ridge Preservation-A Feasibility Study. Clin Oral Implants Res. 2025 Nov 30. doi: 10.1111/clr.70074. Online ahead of print. PMID 41320732